CLINICAL TRIAL: NCT01313663
Title: A Randomized, Open-label, Phase II, 2-arm Multi-center Trial Comparing Maintenance Therapy With Pazopanib or Pemetrexed in Non-progressing Subjects With Metastatic Stage IVA and IVB Non-squamous Non-small Cell Lung Cancer (NSCLC) After Induction Therapy With Carboplatin + Pemetrexed or Cisplatin + Pemetrexed
Brief Title: A Study to Evaluate Pazopanib in Comparison to Pemetrexed in Maintenance Setting in Non-progressing Subjects With Metastatic Stage IVA and IVB Non-squamous Non-small Cell Lung Cancer (NSCLC) Population
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113758
Record Dates: First submitted 2011-01-27; First posted 2011-03-14 (Estimated); Results first posted 2013-04-29 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2013-10

CONDITIONS: Lung Cancer, Small Cell
Keywords: GW786034; non-small cell lung cancer; NSCLC; pemetrexed; pazopanib
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — pazopanib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pazopanib (Experimental): oral agent, administered at 800 mg daily (400 mg tablets x 2). Dose can be reduced, interrupted or discontinued due to adverse events or intolerance
  Interventions: Drug: pazopanib
- Pemetrexed (Active Comparator): pemetrexed IV 500 mg/m2 once every 3 weeks
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pazopanib — oral agent, administered at 800 mg daily (400 mg tablets x 2). Dose can be reduced, interrupted or discontinued due to adverse events or intolerance
  Arms: Pazopanib
Drug: pemetrexed — pemetrexed IV 500 mg/m2 once every 3 weeks
  Arms: Pemetrexed

SUMMARY:
This is a Phase II, randomized, open-label, multi-center study in advanced (Stage IVA and IVB subjects per the International Association for the Study of Lung Cancer (IASLC) 2009 Lung cancer staging schema) non-squamous NSCLC subjects comparing pazopanib relative to pemetrexed in the maintenance setting. Subjects should have completed 4-6 cycles of induction therapy with carboplatin + pemetrexed or cisplatin + pemetrexed and have had Stable Disease (SD), Partial Response (PR) or Complete Response (CR) as the best response to be enrolled into the study. The primary objective is to estimate the hazard ratio of progression free survival (PFS) in advanced NSCLC subjects given maintenance therapy of pazopanib (Arm A) relative to pemetrexed (Arm B). The secondary objectives are: overall survival, response rates, safety and tolerability. A total of approximately 200 subjects will be enrolled and randomized in a 1:1 ratio. Safety and efficacy assessments will be regularly performed on all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed written Informed Consent.
* Subjects must complete 4 to 6 cycles of chemotherapy with carboplatin + pemetrexed or cisplatin + pemetrexed and have had SD, PR or CR at the time of screening/enrolment as the best response.
* Prior surgery and/or localized irradiation for NSCLC is permitted as long as it was a minimum of 4 weeks before entering the study. Subjects with recurrence after previous NSCLC that has been treated with surgery and adjuvant chemotherapy or a radio-chemotherapy regimen with curative intent are eligible, provided 1 year has passed since this treatment ended.
* Histologically or cytologically confirmed diagnosis of predominantly non-squamous cell Stage IVA Wet (with cytology positive Malignant Pleural Effusion (MPE)) or Stage IVB (metastatic) NSCLC.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 12 weeks.
* Must have measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST). A measurable lesion is defined as a lesion that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques, or ≥ 10 mm with spiral computed tomography (CT) scan.
* Able to swallow and retain oral medication.
* Adequate organ system function.
* Women of childbearing potential must have a negative pregnancy test within <= 7 days prior to administration or dispensing of study treatment and agree to use effective contraception.
* Age ≥ 18 years of legal age of consent if different from 18 years.

Exclusion Criteria:

* History of active or any other malignancy other than lung cancer in the 2 yrs prior to the first dose of study drug other than NSCLC. Exception: Subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti- seizure medications for 4 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:
* Active peptic ulcer disease
* Known intraluminal metastatic lesion/s with risk of bleeding
* Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

Malabsorption syndrome Major resection of the stomach or small bowel

* Presence of uncontrolled infection.
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 6 months:

Cardiac angioplasty or stenting Myocardial infarction Unstable angina Coronary artery bypass graft surgery Symptomatic peripheral vascular disease Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).

- Poorly controlled hypertension, defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of

* 90mmHg.

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Blood pressure (BP) must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be <140/90 mmHg in order for a subject to be eligible for the study.

* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti- coagulating agents for at least 6 weeks are eligible.
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
* Evidence of active bleeding or bleeding diathesis.
* Recent hemoptysis (>=½ teaspoon of red blood within 8 weeks before first dose of study drug).
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels (Note: tumor abutting the vessel is acceptable, but contiguous tumor and vessel is not; CT with contrast is strongly recommended to evaluate such lesions).
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that would make the subject inappropriate for study participation including any serious condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Use of any prohibited medication within the timeframes listed in the protocol.
* Prior use of an investigational agent within 28 days or 5 half-lives, whichever is longer, prior the first dose of study drug.
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 (except the value for hemoglobin; see Table 1) and/or that is progressing in severity, except alopecia.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib and/or pemetrexed.
* Inability to interrupt aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs) 2 days before, the day of, and 2 days after the dose of pemetrexed. If a subject is taking an NSAID (COX-2 inhibitors included) or salicylate with a long half-life (e.g.

naproxen, piroxicam, diflusinal, nabumetone, rofecoxib, or celecoxib) it should not be taken 5 days before, the day of, and 2 days after the dose of pemetrexed.

* Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.
* Have clinically significant third-space fluid collections (e.g., ascites or pleural effusions) that cannot be controlled by drainage or other procedures prior to Day 1, Cycle 1.
* Treatment with any of the following anti-cancer therapies:

radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (22):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Ames, Iowa
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Pikeville, Kentucky
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Latham, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Garland, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Mesquite, Texas
  - GSK Investigational Site, San Marcos, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) must have received at least 4-6 cycles of induction therapy with carboplatin + pemetrexed or cisplatin + pemetrexed and should have had stable disease, partial response, or complete response as best response at the time of screening/enrollment. Par. were stratified by disease stage and cycles of induction therapy at enrollment.
Groups:
- Pemetrexed 500 mg/m^2: Participants received an intravenous (IV) infusion of pemetrexed (500 mg per meters squared [mg/m^2]) over 10 minutes on Day 1 of each 21-day cycle. Participants received study treatment until disease progression, death, unacceptable adverse event, withdrawal of consent, or physician decision. Participants who withdrew due to an adverse event or disease progression were followed for survival.
- Pazopanib 800 mg: Participants received pazopanib 800 milligrams (mg) orally once a day at approximately the same time each day, either 1 hour before a meal or 2 hours after a meal. The tablets were to be swallowed whole and were not to be crushed or broken. Participants received study treatment until disease progression, death, unacceptable adverse event, withdrawal of consent, or physician decision. Participants who withdrew due to an adverse event or disease progression were followed for survival.
Period: Overall Study
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Started | 9 | 11
Completed | 5 | 3
Not Completed | 4 | 8
Not completed — Study Closed/Terminated | 2 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.1 (12.09) | 72.6 (11.81) | 72.0 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 9 | 10 | 19
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the interval between the date of randomization and the first documented sign of investigator-assessed (per Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) disease progression (PD) or death, whichever occurs first. The date of documented PD is the date of lesion evaluation in the case of radiological PD and the date of symptomatic cancer progression in the case of symptomatic progression (radiological confirmation is required). PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started. If the participant received subsequent anti-cancer therapy prior to the date of documented progression or death, PFS was to be censored at the last adequate assessment (LAA) prior to the initiation of therapy. Otherwise, if the participant did not have a documented date of progression or death, PFS was to be censored at the date of the LAA.
Time Frame: From randomization until the first documented sign of investigator-assessed disease progression or death, whichever occurred first (average of 10 study weeks)
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to study treatment regardless of whether or not treatment was administered
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 11
weeks | 10.3 [5.3 to NA] — There were too few events of progression/death to calculate the upper limit (UL) of the confidence interval (CI). | 12.7 [6.0 to NA] — There were too few events of progression/death to calculate the upper limit (UL) of the confidence interval (CI).
Statistical Analysis 1: Comparison: Pemetrexed 500 mg/m^2 vs Pazopanib 800 mg; Test type: Superiority or Other; Hazard Ratio (HR) = 0.92, 90% CI 2-sided [0.32 to 2.65] — HRs were estimated using the Pike estimator. The hazard ratio and p-value from the stratified log-rank test were adjusted for disease stage at Baseline only, due to sparse data

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the interval between the date of randomization and the date of death from any cause.
Time Frame: From randomization until disease progression or death (up to Study Week 78)
Population: The study size (20 participants) and follow up were not adequate to assess overall survival. Participants who had not died at the time of the cut-off for the analysis were to be censored at the date the particpant was last known to be alive.
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants (Par.) With the Indicated Best Overall Response
Description: A par. was defined as a responder if s/he sustained a CR (The disappearance of all target lesions. Any pathological lymph node must be less than 10 millimeters [mm] in the short axis) or PR (At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters) that was confirmed after >=28 days. Response was evaluated by an investigator per RECIST, version 1.1. A par. without a post-Baseline assessment was considered a non-responder. Stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started). To qualify as a best response of SD, a response of SD had to be observed >=12 weeks after randomization. A par. who was not evaluable had no scans at all or did not have a confirmatory scan.
Time Frame: From randomization until the time of the first documented evidence of a confirmed complete response (CR) or partial response (PR) (average of 10 weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 11
participants
  CR | 0 | 0
  PR | 0 | 0
  SD | 2 | 2
  PD | 4 | 4
  Not evaluable | 3 | 5

4. Secondary Outcome: Number of Participants With Any Non-serious On-therapy Adverse Event (AE: Occurring in >=5% Participants in Any Treatment Arm) and Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect. In addition, all Grade 4 laboratory abnormalities and other medically important events that require medical or surgical intervention to prevent one of the outcomes listed previously are considered to be SAEs. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the time the first dose of study treatment was administered until 28 days following discontinuation of study treatment regardless of initiation of a new cancer therapy or transfer to hospice (up to Study Week 55)
Population: Safety Population: all participants who were randomized and took at least one dose of study medication. This population was based on the actual treatment received, if it differed from that to which the participant was randomized.
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 10
participants
  Non-serious AEs | 9 | 9
  SAEs | 2 | 2

5. Secondary Outcome: Time on Study Treatment (Pazopanib), as a Measure of Extent of Exposure
Description: Time on study treatment, as a measure of extent of exposure, was assessed in all participants who received pazopanib. Time on study treatment was not measured in participants receiving pemetrexed. For these participants, extent of exposure was measured as the mean number of dosing cycles and dose intensity. See the outcome measures entitled "Mean number of dosing cycles, as a measure of extent of exposure" and "Average dose of pemetrexed for all cycles, as a measure of extent of exposure," respectively, for pemetrexed data.
Time Frame: From the first day to the last day of treatment (average of 8 weeks)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 0 | 10
months |  | 1.8 (1.02)

6. Secondary Outcome: Mean Daily Dose, as a Measure of Extent of Exposure
Description: Mean daily dose, as a measure of extent of exposure, was assessed in all participants who received pazopanib. Mean daily dose was not measured in participants receiving pemetrexed. For these participants, extent of exposure was measured as the mean number of dosing cycles and dose intensity. See the outcome measures entitled "Mean number of dosing cycles, as a measure of extent of exposure" and "Average dose of pemetrexed for all cycles, as a measure of extent of exposure," respectively, for pemetrexed data.
Time Frame: From the first day to the last day of treatment (average of 8 weeks)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 0 | 10
milligrams |  | 751.3 (82.85)

7. Secondary Outcome: Mean Number of Pemetrexed Dosing Cycles, as a Measure of Extent of Exposure
Description: Duration of therapy/time on study treatment, measured as the mean number of pemetrexed dosing cycles as a measure of extent of exposure, was assessed in all participants who received pemetrexed. The mean number of dosing cycles was not measured in participants receiving pazopanib. For these participants, extent of exposure was measured as the time on study treatment and mean daily dose. See the outcome measures entitled "Time on study treatment (pazopanib), as a measure of extent of exposure" and "Mean daily dose, as a measure of extent of exposure," respectively, for pazopanib data.
Time Frame: From the time the first dose of study treatment was administered until discontinuation of the study or death (average of 16 weeks)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: number of cycles
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 0
number of cycles | 5.2 (5.49) |

8. Secondary Outcome: Average Dose of Pemetrexed for All Cycles, as a Measure of Extent of Exposure
Description: The average dose of pemetrexed for all cycles, as a measure of extent of exposure, was assessed in all participants who received pemetrexed. The average dose was not measured in participants receiving pazopanib. For these participants, extent of exposure was measured as the time on study treatment and mean daily dose. See the outcome measures entitled "Time on study treatment (pazopanib), as a measure of extent of exposure" and "Mean daily dose, as a measure of extent of exposure," respectively, for pazopanib data.
Time Frame: as for outcome 7
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milligrams per meters squared (m^2)
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 0
milligrams per meters squared (m^2) | 499.54 (30.222) |

9. Secondary Outcome: Number of Participants With Any AE (Serious or Non-serious) Leading to Withdrawal From Study Treatment
Description: An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect. In addition, all Grade 4 laboratory abnormalities and other medically important events that require medical or surgical intervention to prevent one of the outcomes listed previously are considered to be SAEs. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs. A participant cold have been withdrawn fom study treatment due to an SAE or AE.
Time Frame: From the time the first dose of study treatment was administered until withdrawal from study treatment (up to Study Week 55)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 10
participants | 2 | 2

10. Secondary Outcome: Number of Participants With Any On-therapy AE (Serious or Non-serious) Leading to Dose Reductions (DRs) or Interruptions/Delays in the Study
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect. In addition, all Grade 4 laboratory abnormalities and other medically important events that require medical or surgical intervention to prevent one of the outcomes listed previously are considered to be SAEs. Refer to the general Adverse AE/SAE module for a complete list of AEs/SAEs. Management of AEs may require DRs/interruptions in study treatment. If necessary, the pazopanib dose should be reduced stepwise by 200 mg at each step. DRs for pemetrexed were 50-75% of prior dose based on the toxicity leading to DR.
Time Frame: From the time the first dose of study treatment was administered until discontinuation of treatment (up to Study Week 55)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 10
participants
  Dose reductions | 1 | 2
  Dose interruptions/delays | 1 | 3

11. Secondary Outcome: Number of Participants With the Indicated Worst-case Change From Baseline in Blood Pressure
Description: Systolic and diastolic blood pressure (BP) were measured. Categories correspond to the following Common Terminology Criteria for Adverse Events (CTCAE) grades: normal, <120/80 millimeters of mercury (mmHg); prehypertension, 120-139/80-89 mmHg, warranting intervention in participants with high risk; stage I hypertension, 140-159/90-99 mmHg, warranting intervention; and stage II hypertension >/=160/100, warranting immediate attentive intervention to prevent acute symptoms. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Participants with a missing Baseline value were assumed to have a Baseline value of <120 for systolic BP (SBP) and <80 for diastolic BP (DBP).
Time Frame: From the time of the first dose of study treatment until 28 days following discontinuation of study treatment (up to Study Week 55)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 10
participants
  SBP, increase to 120-139 mmHg | 2 | 1
  SBP, increase to 140-159 mmHg | 3 | 3
  SBP, increase to >=160 mmHg | 1 | 4
  DBP, increase to 80-89 mmHg | 2 | 3
  DBP, increase to 90-99 mmHg | 1 | 5
  DBP, increase to >=100 mmHg | 0 | 0

12. Secondary Outcome: Number of Participants With a Increase From Baseline in Bazett's QTc at the Indicated Time Points
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. In clinical studies with pazopanib, events of QT prolongation have occurred.
Time Frame: Baseline; Week 6; Week 15; every 9 weeks in the first 6 months; every 12 weeks in the next 6 months; and, after 1 year, every 6 months (up to Study Week 55)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 10
participants | 0 | 0

13. Secondary Outcome: Number of Participants With a Change From Baseline Grade to Grade 3 and 4 for the Indicated Clinical Laboratory Parameters
Description: Hematology and clinical chemistry data were summarized according to National Cancer Institutes (NCI) CTCAE grade, version 4.0. Grade 1, Mild; Grade 2, Moderate; Grade 3, Severe; Grade 4, Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to Grade 3 or Grade 4 occurred. Participants with missing Baseline grades were assumed to have a Baseline grade of 0. Lymphocyte count increased: Grade 3, <500 - 200/millimeters cubed (mm^3); <0.5 - 0.2x 10e9/Liters (L); Grade 4, <200/mm^3; <0.2x 10e9/L. Lymphocyte count decreased: Grade 3, >20000/mm^3; Grade 4, NA. Hyperglycemia; Grade 3, >250 - 500 milligrams per deciliter (mg/dL); >13.9 - 27.8 millimoles per Liter (mmol/L); hospitalization indicated; Grade 4, >500 mg/dL; >27.8 mmol/L; life-threatening consequences. Hypophosphatemia (inorganic phosphorus): Grade 3, <2.0 - 1.0 mg/dL, <0.6 - 0.3 mmol/L; Grade 4, <1.0 mg/dL, <0.3 mmol/L, life-threatening consequences.
Time Frame: as for outcome 11
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 10
participants
  Lymphocytes, Grade 3 | 2 | 1
  Hyperglycemia, Grade 3 | 0 | 1
  Phosphorus inorganic, Grade 3 | 0 | 1

14. Secondary Outcome: Number of Participants With the Indicated Grade Changes From Baseline Grade in Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (Alk. Phos.), and Total Bilirubin (TB)
Description: The laboratory parameters AST, ALT, Alk. Phos., and TB were summarized according to NCI CTCAE grade, version 4.0. Grade 1, Mild; Grade 2, Moderate; Grade 3, Severe; Grade 4, Life-threatening or disabling; Grade 5, Death. Data are presented for any grade increase, increase to Grade 3, and increase to Grade 4. Participants with missing Baseline grades were assumed to have a Baseline grade of 0. AST/ALT: Grade 1, >upper limit of normal (ULN) - 3.0x ULN; Grade 2, >3.0 to 5.0x ULN; Grade 3, >5.0 - 20.0x ULN; Grade 4, >20.0x ULN; Grade 5, not available (NA). Alk. Phos.: Grade 1, >ULN - 2.5x ULN; Grade 2, >2.5 - 5.0x ULN; Grade 3, >5.0 - 20.0x ULN; Grade 4, >20.0x ULN; Grade 5, NA. TB: Grade 1, >ULN - >1.5x ULN; Grade 2, >1.5 - 3.0x ULN; Grade 3, >3.0 - 10.0x ULN; Grade 4, >10.0x ULN; Grade 5, NA.
Time Frame: as for outcome 11
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 10
participants
  AST, any Grade | 1 | 0
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 0 | 0
  ALT, any Grade | 1 | 1
  ALT, Grade 3 | 0 | 0
  ALT, Grade 4 | 0 | 0
  Alk. Phos., any Grade | 0 | 1
  Alk. Phos., Grade 3 | 0 | 0
  Alk. Phos., Grade 4 | 0 | 0
  TB, any Grade | 0 | 0
  TB, Grade 3 | 0 | 0
  TB, Grade 4 | 0 | 0

15. Secondary Outcome: Number of Participants With the Indicated Changes From Baseline Value in Lactate Dehydrogenase (LDH)
Description: Change from Baseline in the laboratory parameter LDH was assessed as "decrease to low," "change to normal" of "no change," and "increase to high." Participants with missing Baseline values were assumed to have a normal Baseline value. There is no standard normal range for LDH.
Time Frame: as for outcome 11
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Number analyzed (Participants) | 9 | 10
participants
  Decrease to low | 0 | 0
  Change to normal/No change | 4 | 7
  Increase to high | 5 | 3

ADVERSE EVENTS:
Time Frame: Participants were analyzed from the time the first dose of study treatment was administered until 28 days following discontinuation of study treatment regardless of initiation of a new cancer therapy or transfer to hospice (up to Study Week 55).
Description: Serious adverse events (SAEs) and non-serious AEs were collected in the Safety Population, comprisedof all participants who were randomized and took at least one dose of study medication. This population was based on the actual treatment received, if it differed from that to which the participant was randomized.
Arm/Group | Pemetrexed 500 mg/m^2 | Pazopanib 800 mg
Serious Adverse Events (participants affected / at risk) | 2/9 | 2/10
Other Adverse Events (participants affected / at risk) | 9/9 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed 500 mg/m^2 (N=9) | Pazopanib 800 mg (N=10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed 500 mg/m^2 (N=9) | Pazopanib 800 mg (N=10)
Fatigue (General disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 2 | 3
Alanine aminotransferase increased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Headache (Nervous system disorders) | 1 | 2
Hypertension (Vascular disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Upper-airway cough syndrome (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Chills (General disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Malaise (General disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Spinal pain (General disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.